CLINICAL TRIAL: NCT05103033
Title: Systems Analysis and Improvement Approach to Optimize the Task-shared Mental Health Treatment Cascade (SAIA-MH): A Cluster Randomized Trial
Brief Title: Systems Analysis and Improvement Approach to Optimize the Task-shared Mental Health Treatment Cascade (SAIA-MH)
Acronym: SAIA-MH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Comité para a Saúde de Moçambique (Unknown); Ministry of Health, Mozambique (Other Government)
Responsible Party: Principal Investigator, Bradley Wagenaar, Assistant Professor, School of Public Health: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00012527; 1R01MH123682-01A1 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Disorder
Keywords: Outpatient primary care
MeSH Terms: conditions — Mental Disorders | interventions — Mental Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systems Analysis and Improvement Approach (SAIA) for mental health (Experimental): Those receiving SAIA-MH will attend a 1-week in-person training for facility learning collaboratives. Following the 1-week in-person training, SAIA-MH standard operating procedures will be implemented, including: (1) structured internal/external facilitation following tablet-based guides used in pilot study (1x per week first month; 2x per week for next two months; 1x per month for remainder); (2) facilitation in the 5-step SAIA-MH improvement process.
  Interventions: Behavioral: Systems Analysis and Improvement Approach for Mental Health (SAIA-MH)
- Attentional Placebo Control (Other): Control facilities will mimic activities of the intervention group in time and contacts, but without the "active ingredient" of the SAIA-MH implementation strategy
  Interventions: Behavioral: Attentional Placebo Control

INTERVENTIONS:
Behavioral: Systems Analysis and Improvement Approach for Mental Health (SAIA-MH) — The 5 steps of SAIA-MH include: (1) cascade analysis to visualize treatment cascade drop-offs and prioritize areas for system improvements; (2) process mapping to identify modifiable facility-level bottlenecks; (3) identification and implementation of modifications to improve system performance; (4) assessment of modification effects on the cascade; and (5) repeated analysis and improvement cycles.
  Arms: Systems Analysis and Improvement Approach (SAIA) for mental health
Behavioral: Attentional Placebo Control — Facilities randomized to attentional placebo control will attend a 1-week in-person training which will include the same minimum staff above for SAIA-MH. This training will focus on reviewing data collection tools, ethics, mental health stigma and burnout for mental health professionals. Following the 1-week in person training, attentional placebo control facilities will receive regular supervision following the same schedule as SAIA-MH focused on reviewing data collection tools.
  Arms: Attentional Placebo Control

SUMMARY:
The purpose of this study is to test the effectiveness of a multicomponent implementation strategy entitled the Systems Analysis and Improvement Approach for mental health (SAIA-M) using a cluster randomized trial at the health facility level. SAIA-MH focuses on improving the mental health treatment cascade in primary outpatient mental healthcare. The mental health treatment cascade is a model that outlines the sequential, linked treatment steps that people with mental illness must navigate, from initial diagnosis to symptom/function improvement.

This study will also assess the potential mechanisms by which the SAIA-MH implementation strategy works, or does not work, along with the cost and effectiveness of scaling-up SAIA-MH in Mozambique.

DETAILED DESCRIPTION:
Due to a shortage of 1.2 million mental health (MH) workers across low- and middle-income countries (LMICs), academic and policy leaders have advocated scaling-up task-sharing to lower-level providers to close the mental health care gap, which exceeds 90% in many LMICs. While task-sharing may increase access to care, limited attention has been paid to quality of care provided by lower-level providers. Task-shared outpatient management of mental health in Mozambique has shown low rates of retention in care (40%), medication adherence (<15%), and proportion of patients achieving function improvement (<5%). Similarly high rates of loss-to-follow-up, poor adherence, and poor patient outcomes have been reported across other LMICs. To our knowledge, there are no evidence-based implementation strategies targeting optimization of the MH treatment cascade in low-resource settings. This is an urgent need for the field of MH care delivery globally.

The MH treatment cascade is a model that outlines the sequential, linked treatment steps that people with mental illness must navigate, from initial diagnosis to symptom/function improvement. Quality problems in one step of a treatment cascade can have non-linear and compounding impacts across the larger complex care system. Implementation strategies focused on only one step in a cascade can potentially contribute to unintended system bottlenecks and quality of care issues. By contrast, the "Systems Analysis and Improvement Approach (SAIA)" is a multicomponent implementation strategy focused on optimizing an entire treatment cascade. SAIA blends facilitation, enhanced local clinical consultation, and the creation of facility-level learning collaboratives with systems-engineering tools in a 5-step approach specifically developed for task-shared providers, which include: (1) cascade analysis to visualize treatment cascade drop-offs and prioritize areas for system improvements; (2) process mapping to identify modifiable facility-level bottlenecks; (3) identification and implementation of modifications to improve system performance; (4) assessment of modification effects on the cascade; and (5) repeated analysis and improvement cycles. A previous cluster RCT established effectiveness of SAIA for HIV treatment cascade improvement (R01HD075057; PI: Sherr). However, no effectiveness data exist on SAIA applied to other complex treatment cascades - such as task-shared MH care. Preliminary data suggest that applying SAIA to MH treatment cascade optimization (SAIA-MH; R21MH113691; PI: Wagenaar) is feasible, acceptable, and can result in clinically-significant treatment cascade improvements; Five months of SAIA-MH implementation resulted in a 1.5-fold increase in medication adherence (aOR: 1.5; CI: 1.2, 1.9) and a 3.7-fold increase in function improvement (aOR: 3.7; CI: 2.5, 5.4). These data suggest that SAIA-MH is a promising strategy for task-shared MH systems improvement globally. Our specific aims are to:

Primary Aim 1: Test the effectiveness of the SAIA-MH strategy using a pragmatic cluster RCT design and assess determinants of implementation success. The investigators will implement SAIA-MH using a 3-year parallel cluster RCT across 8 intervention and 8 attentional control facilities and evaluate effects on mental health function improvement (primary) and retention / medication adherence (secondary). Two years of study implementation will be followed by a 1-year maintenance phase to examine routine fidelity and sustainability. The Consolidated Framework for Implementation Research (CFIR) will be used to assess determinants of implementation success.

Secondary Aim 1: Test causal pathway models to analyze mechanisms of action for effects (or non-effects) of the SAIA-MH implementation strategy. Using 3-years of monthly data on strategy-mechanism linkages, moderators, preconditions, and outcomes for the full 8 intervention and 8 attentional control facilities, the investigators will examine causal pathway effect estimates using longitudinal structural equation modeling. Qualitative CFIR data from Primary Aim 1 will contextualize quantitative path analyses.

Specific Aim 2: Estimate the cost and cost-effectiveness of scaling-up SAIA-MH in Mozambique. The investigators will conduct micro-costing and time-and-motion observation of the SAIA-MH RCT to estimate costs of implementing the intervention. The investigators will construct a Markov model parameterized with cost and outcome data from the SAIA-MH RCT to project budget impact and cost-effectiveness for SAIA-MH scale-up to provincial and national levels.

ELIGIBILITY:
Inclusion Criteria for Primary and Secondary Outcomes:

1. Patient diagnosed with a mental health condition in outpatient primary care, prescribed a medication, and given a follow-up date.

Exclusion Criteria for Primary and Secondary Outcomes:

1. Patient enrolled in treatment outside of targeted mental health systems analysis and improvement approach (SAIA-MH) facilities.
2. Patients not prescribed a medication.
3. Patients not given a follow-up date.

Inclusion Criteria for Qualitative Interviews:

1. Mental health workers currently working and collaborating on the treatment of outpatient mental health patients in target clinics in Sofala or Manica provinces, Mozambique.
2. Mental health workers must be employed by Ministry of Health.
3. Mental health managers or directors currently supervising mental health workers who are leading treatment of outpatient mental health patients in target clinics in Sofala or Manica provinces, Mozambique. Must be employed by the Ministry of Health.

Exclusion Criteria for Qualitative Interviews:

1. Health worker not involved in outpatient mental healthcare delivery. Health worker not employed by the Ministry of Health.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient Function Improvement | data collection will occur over 6 months baseline, 24-month intervention and 12-month sustainment period
  Patient function improvement is evaluated for all patients diagnosed with a mental disorder, prescribed a medication, given a follow-up date, and who return at least once. All patients diagnosed with a mental disorder in target clinics will have function improvement measured by the WHODAS 2.0 at each clinic visit.
  Improvement will be determined as patients with at least 1 follow-up visits who score less than 10 on the WHODAS 2.0 or have a 50% reduction in their baseline WHODAS 2.0 score.

SECONDARY OUTCOMES:
Patient Retention | data collection will occur over 6 months baseline, 24-month intervention and 12-month sustainment period
  Patient retention is evaluated for all patients diagnosed with a mental disorder, prescribed a medication, given a follow-up date, and who return at least once. This outcome evaluates whether these individuals returned for their scheduled follow-up visit in less than or equal to 30 days.
Patient Medication Adherence | data collection will occur over 6 months baseline, 24-month intervention and 12-month sustainment period
  Medication adherence is evaluated for all patients diagnosed with a mental disorder, prescribed a medication, given a follow-up date, and who return at least once. These patients are considered to have potentially achieved medication adherence if they return for their follow-up visit and medication refill in less days than they had pills dispensed at their previous visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Wagenaar, MPH, PhD, Principal Investigator — University of Washington
Locations (16):
- Mozambique (16):
  - District Hospital Catandica, Catandica, Manica Province
  - Urban Health Center Nhamaonha, Chimoio, Manica Province
  - Urban Health Center Vila Nova, Chimoio, Manica Province
  - District Hospital Gondola, Gondola, Manica Province
  - Rural Health Center Macate, Macate, Manica Province
  - Rural Health Center Sussundenga Sede, Sussundenga, Manica Province
  - Rural Health Center Vanduzi, Vanduzi, Manica Province
  - Urban Health Center Chingussura, Beira, Sofala
  - Urban Health Center Inhamizua, Beira, Sofala
  - Urban Health Center Macurungo, Beira, Sofala
  - Urban Health Center Mascarenhas, Beira, Sofala
  - Hospital Muxúngue, Chibabava, Sofala
  - Rural Health Center Mafambisse, Dondo, Sofala
  - Urban Health Center Dondo Sede, Dondo, Sofala
  - Rural Hospital Nhamatanda, Nhamatanda, Sofala
  - District Hospital Manica, Manica

REFERENCES:
- [Derived] Turner M, Muanido A, Cumbe V, Jala JN Jr, Armando EE, Mambuque E Jr, Faduque F, Xerinda ER, Sherr K, Weiner BJ, Flaherty BP, Sharma M, Wagenaar BH. Mental health care cascade performance and associated factors: longitudinal analyses of routine Ministry of Health services in Mozambique. BMJ Public Health. 2025 Mar 13;3(1):e001024. doi: 10.1136/bmjph-2024-001024. eCollection 2025. PMID 40099137
- [Derived] Cumbe VFJ, Muanido AG, Turner M, Ramiro I, Sherr K, Weiner BJ, Flaherty BP, Sharma M, Faduque F, Xerinda ER, Wagenaar BH. Systems analysis and improvement approach to optimize outpatient mental health treatment cascades in Mozambique (SAIA-MH): study protocol for a cluster randomized trial. Implement Sci. 2022 Jun 6;17(1):37. doi: 10.1186/s13012-022-01213-8. PMID 35668423